CLINICAL TRIAL: NCT01722110
Title: A Randomized, Balanced, Open Label, Two Treatment, Two Period, Two Sequence, Single Dose, Crossover, Bioequivalence Study of Indomethacin Extended-Release Capsules 75 mg of Ipca Laboratories Ltd., With Indomethacin Extended-Release Capsules USP 75 mg of Epic Pharma, USA, in Normal, Healthy, Adult, Male and Female Human Subjects Under Fed Conditions.
Brief Title: Bioequivalence Study of Indomethacin Extended-Release Capsules 75 mg Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IPCA Laboratories Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Ipca/ARL-10/436
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indomethacin Extended-Release Capsules USP 75 mg (Experimental): Indomethacin Extended-Release Capsules USP 75 mg of Ipca Laboratories Limited, India
  Interventions: Drug: Indomethacin Extended-Release Capsules USP 75 mg
- Indomethacin Extended Release Capsules USP 75 mg (Active Comparator): Indomethacin Extended Release Capsules USP 75 mg of Epic Pharma, USA.
  Interventions: Drug: Indomethacin Extended Release Capsules USP 75 mg

INTERVENTIONS:
Drug: Indomethacin Extended-Release Capsules USP 75 mg — 75 mg tablet once a day
  Other Names: Test Product
  Arms: Indomethacin Extended-Release Capsules USP 75 mg
Drug: Indomethacin Extended Release Capsules USP 75 mg — 75 mg tablet once a day
  Arms: Indomethacin Extended Release Capsules USP 75 mg

SUMMARY:
This is a randomized, balanced, open Label, two-treatment, two-period, two-sequence, single dose, crossover pivotal study. The purpose of this study is to assess the bioequivalence between Test Product and the corresponding Reference Product under fed condition in normal, healthy, adult, male and female human subjects.

DETAILED DESCRIPTION:
Objective of this pivotal study was to assess the bioequivalence between Test Product: Indomethacin Extended-Release Capsules USP 75 mg of Ipca Laboratories Limited, India and the corresponding Reference Product: Indomethacin Extended-Release Capsules USP 75 mg of Epic Pharma, USA, under fed condition in normal, healthy, adult, male and female human subjects in a randomized crossover study.

The study was conducted with 32 healthy adult subjects. In each study period, a single 75 mg dose of either test or reference was administered to the subjects as per the randomization schedule in each study period with about 240 mL of water at ambient temperature in sitting position.

The duration of the clinical phase was approximately 10 days including washout period of at least 7 days between administrations of study drug in each study period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non pregnant female human subjects, age in the range of 18 - 45 years.
2. Body weight within ± 15% of ideal weight as related to height and body frame according to Life Insurance Corporation (LIC) Chart.
3. Subjects with normal findings as determined by baseline history, physical examination and vital sign examination (blood pressure, pulse rate, respiration rate and axillary temperature).
4. Subjects with clinically acceptable findings as determined by haemogram, biochemistry, urinalysis and 12 lead ECG.
5. Subject's willing to give written informed consent.
6. Willingness to follow the protocol requirements especially abstaining from xanthine containing food or beverages (chocolates, tea, coffee or cola drinks) or grapefruit juice, any alcoholic products, the use of cigarettes and tobacco products for 48 hours prior to dosing until after the last blood sample collection in each study period and adherence to food, fluid and posture restrictions.
7. No history of significant alcoholism.
8. No history of drug abuse (benzodiazepines and barbiturates) for the last one month and other illegal drugs for the last 6 months.
9. Non-smokers were included.

Exclusion Criteria:

1. Known history of hypersensitivity to Indomethacin or related drugs.
2. Requiring medication for any ailment having enzyme-modifying activity in the previous 28 days, prior to dosing day.
3. Subjects who have taken prescription medications or over-the-counter products (including vitamins and minerals) within 14 days prior to administration of Investigational Product.
4. Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract, blood-forming organs etc.
5. History of cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic, haematological, gastrointestinal, endocrine, immunological or psychiatric diseases.
6. Participation in a clinical drug study or bioequivalence study 90 days prior to present study.
7. History of malignancy or other serious diseases.
8. Blood donation 90 days prior to the commencement of the study.
9. Subjects with positive HIV tests, HBsAg or Hepatitis-C tests.
10. Found positive in breath alcohol test.
11. Found positive in urine test for drug abuse.
12. History of problem in swallowing.
13. Any contraindication to blood sampling.
14. Found positive serum Beta- hCG (Human Chorionic Gonadotropin) test.
15. Lactating women (currently breast feeding).
16. Female subjects not confirming to using birth control measures, from the date of screening until the completion of the study. Abstinence, barrier methods (condom, diaphragm, etc.) were acceptable. Use of hormonal contraceptives either oral or implants.
17. Female subjects whose menstruation cycle coincided with the study periods.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Bioequivalence is based on Cmax and AUC parameters. | 2 months
  Sampling Hours: Pre-dose and at 0.50, 1.00, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 6.00, 7.00, 8.00, 9.00, 10.00, 12.00, 16.00, 20.00, 24.00, 36.00 and 48.00 hrs post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Suhas Khandave, M.D., Principal Investigator — Accutest Research Lab (I) Pvt. Ltd.
Locations (1):
- Accutest Research Lab (I) Pvt. Ltd., Navi Mumbai, Maharashtra, India